CLINICAL TRIAL: NCT07168122
Title: Study for Reference Intervals and Optimal Cut-offs for Salivary Cortisol
Brief Title: Establishment and Clinical Application of Reference Intervals of Salivary Cortisol
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Principal Investigator, Professor, Chief Physician, Deputy Director, Shanghai 6th People's Hospital
Other Study IDs: 20250811
Record Dates: First submitted 2025-08-27; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Healthy Adult; Cushing Syndrome; Adrenal Insufficiency
MeSH Terms: conditions — Cushing Syndrome; Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (3):
- Heathy Volunteers: 120 Healthy Volunteers for the establishment of reference intervals of salivary cortisol
- Cushing's sydrome: 50 cases diagnosed with Cushing's sydrome
- Adrenal insufficiency: 50 cases diagnosed with adrenal insufficiency

SUMMARY:
The goal of this observational study is to establish the normal reference intervals of salivary cortisol and optimal cut-offs for Cushing's sydrome and adrenal insufficiency.

DETAILED DESCRIPTION:
Saliva testing is a non-invasive alternative to blood tests for measuring cortisol, a key hormone for assessing endocrine status and diagnosing conditions like Cushing's syndrome. It accurately reflects physiologically active free cortisol. However, its clinical use is hampered by extremely low cortisol concentrations and the lack of reliable detection methods. We have developed two advanced technologies: an immunomagnetic-bead-based LC-MS assay with simplified preparation, and a fluorescence immunoassay system for point-of-care testing. To promote their clinical adoption, this study will establish normal reference intervals of salivary cortisol for both methods in a healthy population and optimal cut-offs in cases of Cushing's sydrome and adrenal insufficiency.

ELIGIBILITY:
Healthy Volunteers:

Inclusion Criteria:

1. Age ≥ 18 and ≤ 60 years old;
2. Body mass index (BMI) ≥ 18.5 and ≤ 24.9 kg*m^-2;
3. No previous history of chronic diseases such as hyperglycemia, hypertension, dyslipidemia, coronary heart disease and stroke;
4. Normal glucose regulation, defined as: fasting blood-glucose < 5.6 mmol/L, 2-hour blood-glucose after glucose load < 7.8 mmol/L, and glycated hemoglobin (HbA1c) < 5.7%.

Exclusion Criteria:

1. Liver or kidney dysfunction, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or direct bilirubin higher than 1.5 times the upper limit of normal, or serum creatinine >115 μmol/L;
2. Pregnancy or lactation women, or people with cancer or mental illness;
3. Factors affecting cortisol levels, including hypothalamus-pituitary-adrenal axis disease, autoimmune disease (systemic lupus erythematosus, rheumatoid arthritis, etc.), diagnosed mental disease, Alzheimer's disease, alcoholism (alcohol > 60 g/d for male, >40 g/d for women) and corticosteroid therapy in the past 3 months (females with contraceptives or estrogen);
4. Factors affecting saliva collection, such as serious oral problems (oral ulcers, gingival bleeding);
5. Night shift workers, who are awake from 11:00 PM to 7:00 AM;
6. Acute infection (body temperature ≥ 37.3 ℃ or C-reactive protein > 50 mg/L).

Cases:

Inclusion Criteria:

1. Aged 18 to 80 years old;
2. Patients with suspected Cushing's syndrome or adrenal insufficiency.

Exclusion Criteria:

1. Corticosteroid therapy within the last 6 weeks;
2. Acute infection;
3. Severe oral conditions;
4. Severe liver and kidney dysfunction;
5. Alcoholism, depression, or other psychiatric disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants are enrolled from Shanghai Sixth People's Hospital, Shanghai.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Reference intervals of salivary cortisol | 8:00, 16:00 and 23:00 on the day of sample collection
  Salivary cortisol levels were evaluated by immunomagnetic-bead-based LC-MS assay and fluorescence immunoassay system to establish its reference intervals according to the 2.5th and 97.5th percentiles.
Optimal cut-off and diagnostic accuracy of salivary cortisol in Cushing's syndrome | 23:00 on the day of sample collection
  The diagnostic cut-off for each analysis method was defined as either the calculated upper reference interval (97.5th percentile) or the optimal value determined by the Youden index. The sensitivity, specificity and area under curve for Cushing's syndrome was calculated using samples from all available healthy controls and cases.
Optimal cut-off and diagnostic accuracy of salivary cortisol in adrenal insufficiency | 8:00 on the day of sample collection
  The diagnostic cut-off for each analysis method was defined as either the calculated lower reference intervals (2.5th percentile) or the optimal value determined by the Youden index. The sensitivity, specificity and area under curve for adrenal insufficiency was calculated using samples from all available healthy controls and cases.
Comparison of diagnostic accuracy of salivary cortisol in Cushing's syndrome and adrenal insufficiency | 8:00 or 23:00 on the day of sample collection
  The diagnostic accuracies of the fluorescence immunoassay system and the immunomagnetic-bead-based LC-MS assay were compared by analyzing their areas under the receiver operating characteristic (ROC) curves using DeLong's test for paired statistics.

SECONDARY OUTCOMES:
Agreement in assessment of salivary cortisol | 8:00, 16:00 and 23:00 on the day of sample collection
  To assess the agreement in assessment of salivary cortisol between immunomagnetic-bead-based LC-MS assay and fluorescence immunoassay system
Between-groups differences in salivary cortisol of healthy volunteers with different age ranges | 8:00, 16:00 and 23:00 on the day of sample collection
  Comparsion of salivary cortisol levels in subgroups of age
Between-groups differences in salivary cortisol of healthy volunteers with different sex | 8:00, 16:00 and 23:00 on the day of sample collection
  Comparsion of salivary cortisol levels in subgroups of sex
Between-groups differences in salivary cortisol of healthy volunteers with different body mass index ranges | 8:00, 16:00 and 23:00 on the day of sample collection
  Comparsion of salivary cortisol levels in subgroups of body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No